CLINICAL TRIAL: NCT02317991
Title: Phase II Study of Nab-Paclitaxel and Ramucirumab for the Second-line Treatment of Patients With Metastatic Gastroesophageal Cancer
Brief Title: Study of Nab-Paclitaxel and Ramucirumab as Second-line Treatment for Patients With Metastatic Gastroesophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 201
Record Dates: First submitted 2014-12-09; First posted 2014-12-17 (Estimated); Results first posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Gastroesophageal Cancer
Keywords: gastroesophageal adenocarcinoma; nab-paclitaxel; Abraxane; ramucirumab; Cyramza; GE junction
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- nab-paclitaxel and ramucirumab (Experimental): All patients will receive 125 mg/m^2 of nab-Paclitaxel intravenously (IV) on Days 1, 8, and 15 of a 28-day cycle (weekly for 3 weeks, with 1 week of rest).
  Patients will receive ramucirumab 8mg/kg IV in combination with nab-paclitaxel on Days 1 and 15 of the 28-day cycle.
  Interventions: Drug: nab-paclitaxel; Biological: ramucirumab

INTERVENTIONS:
Drug: nab-paclitaxel — nab-paclitaxel 125 mg/m^2 IV
  Other Names: Abraxane; ABI-007
Biological: ramucirumab — Ramucirumab 8 mg/kg IV
  Other Names: Cyramza; IMC-1121B

SUMMARY:
The purpose of this study is to determine whether nab-Paclitaxel (Abraxane®) and ramucirumab (Cyramza®) are effective when used in combination for treating patients with metastatic gastroesophageal cancer who have either progressed or not responded to prior therapy.

DETAILED DESCRIPTION:
Adenocarcinoma of the esophagus and the gastroesophageal junction (GE junction) is the ninth most common cancer worldwide. Ramucirumab (Cyramza®), a monoclonal antibody, is approved as a single agent and in combination with paclitaxel as a treatment for patients with metastatic gastric or GE junction adenocarcinoma whose cancer has progressed after prior chemotherapy. Nab-paclitaxel (Abraxane®) is an albumin-based formulation of paclitaxel which was developed to improve the therapeutic index and reduce toxicity. Nab-paclitaxel is approved in over 40 countries/regions for treatment of various metastatic cancers including breast cancer, non-small cell lung cancer (NSCLC), and pancreatic cancer. In this Phase II study, the investigators propose to combine the less toxic nab-paclitaxel to increase tumor uptake of the drug and improve efficacy while minimizing side effects. The biological rationale of using this combination is that ramucirumab will inhibit tumor angiogenesis and nab-paclitaxel will induce apoptosis of the rapidly dividing tumor cell.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed metastatic adenocarcinoma of the esophagus, GE junction, or stomach who progressed on one prior line of chemotherapy in the metastatic setting.
2. Measurable disease as measured by Response Evaluation Criteria in Solid Tumors (RECIST) criteria Version 1.1.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
4. Adequate hematologic, renal, and hepatic functions
5. Patients must have < Grade 2 pre-existing peripheral neuropathy (per National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v 4.03)
6. Life expectancy > 3 months

Exclusion Criteria:

1. Patients who have received any other investigational agents, chemotherapy, biologic therapy, or radiation therapy within the 28 days prior to Day 1 of the study. For investigational, chemotherapy, or biologic therapy, patients will be allowed on study if five half-lives or greater have elapsed since last dose of drug or 28 days, whichever is shorter.
2. Patients with prior taxane chemotherapy or agents which act by primary anti-angiogenic mechanisms.
3. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit safety or compliance with study requirements or may interfere with the interpretation of the results.
4. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study initiation, or anticipation of need for major surgical procedure during the course of the study.
5. Evidence or history of uncontrolled hypertension, proteinuria, non-healing wound, ulcer, bone fracture, hemoptysis, valvular disease, abdominal fistula, GI perforation, intra-abdominal abscess, bleeding diathesis or coagulopathy that would exclude patients from treatment with anti-angiogenesis agents.
6. Therapeutic anticoagulation with coumarin-derivatives will not be permitted. However, a maximum daily dose of 1 mg will be permitted for port line patency. Anticoagulation with low molecular weight heparin or anti-Factor Xa agents will be allowed.
7. Patients with other concurrent severe and/or uncontrolled medical disease which could compromise safety of treatment as so judged by treating physician (i.e., severely impaired lung function, severe infection, ventricular arrhythmias active ischemic heart disease, known active vasculitis of any cause, chronic liver or renal disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Spigel, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (11):
- United States (11):
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Florida Cancer Specialists-South, Fort Myers, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Florida Cancer Specialists-North, St. Petersburg, Florida
  - Ingalls Cancer Research Center, Harvey, Illinois
  - Research Medical Center, Kansas City, Missouri
  - Oncology Hematology Care, Cincinnati, Ohio
  - Spartanburg Medical Center/Gibbs Cancer Center, Spartanburg, South Carolina
  - Tennessee Oncology, Chattanooga, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Center for Cancer and Blood Disorders, Fort Worth, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Nab-paclitaxel and Ramucirumab: All patients will receive 125 mg/m^2 of nab-Paclitaxel intravenously (IV) on Days 1, 8, and 15 of a 28-day cycle (weekly for 3 weeks, with 1 week of rest).
  Patients will receive ramucirumab 8mg/kg IV in combination with nab-paclitaxel on Days 1 and 15 of the 28-day cycle.
  nab-paclitaxel: nab-paclitaxel 125 mg/m^2 IV
  ramucirumab: Ramucirumab 8 mg/kg IV
Period: Overall Study
Arm/Group | Nab-paclitaxel and Ramucirumab
Started | 65
Completed | 0
Not Completed | 65
Not completed — Adverse Event | 12
Not completed — Death | 4
Not completed — Withdrawal by Subject | 8
Not completed — Progressive Disease | 41

BASELINE CHARACTERISTICS:
Arm/Group | Nab-paclitaxel and Ramucirumab
Number analyzed (Participants) | 65
Age, Continuous [Median (Full Range); unit: years] | 63 [35 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 58
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65
Participants with HER2 positive status (confirmed by FISH) [Count of Participants; unit: Participants] | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Measured from Day 1 of study drug administration to disease progression as defined by Response Evaluation in Solid Tumors Criteria (RECIST v1.1), or death on study from any cause. Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Participants who are alive and free from disease progression were censored at the date of the last adequate tumor assessment. If no adequate post-treatment tumor assessments were obtained for participants, PFS will be censored on Day 1.
Time Frame: up to 1 year
Population: Full analysis set. All enrolled patients who have received at least one dose of study treatment and have a baseline tumor assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-paclitaxel and Ramucirumab
Number analyzed (Participants) | 65
months | 3.8 [3.4 to 5.7]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of patients with confirmed complete response (CR) or confirmed partial response (PR), i.e., two CRs and/or PRs at least 4 weeks apart, according to the RECIST v1.1 criteria. CR=disappearance of all target lesions. PR=at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: every 8 weeks up to 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nab-paclitaxel and Ramucirumab
Number analyzed (Participants) | 65
percentage of participants | 20 [10.3 to 29.7]

3. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the time from the first day of study drug administration (Day 1) to objective disease progression as defined by the RECIST v1.1 criteria. Patients who are alive and free from disease progression will be censored at the date of the last adequate tumor assessment. If no adequate post-treatment tumor assessments were obtained for a patient, TTP will be censored on Day 1. Progressive Disease (PD): At least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or unequivocal progression of non-target lesions or the appearance of one or more new lesions.
Time Frame: up to 1 year
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-paclitaxel and Ramucirumab
Number analyzed (Participants) | 65
months | 4.5 [3.5 to 6.4]

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the first treatment until date of death due to any cause. In the absence of confirmation of death or lack of data beyond follow-up period, the survival time was censored to last date the participant was known to be alive.
Time Frame: up to 1 year
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-paclitaxel and Ramucirumab
Number analyzed (Participants) | 65
months | 8 [6.4 to 10.5]

5. Other Pre Specified Outcome: Number of Participants With Treatment-emergent Adverse Events as a Measure of Safety and Tolerability
Description: Adverse events will be graded utilizing the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03
Time Frame: For duration of treatment, up to of 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-paclitaxel and Ramucirumab
Number analyzed (Participants) | 65
Participants | 62

ADVERSE EVENTS:
Time Frame: For the duration of study treatment, up to 6 months for Serious Adverse Events and Other Adverse Events. Until study follow-up discontinuation, an average of 1 year for All-Cause Mortality.
Description: All patients who received at least one dose of protocol treatment were followed for safety. Adverse events and serious adverse events were collected from the day of the first dose to 30 days after the last dose of the study medication and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03
Arm/Group | Nab-paclitaxel and Ramucirumab
All-Cause Mortality (participants affected / at risk) | 51/65
Serious Adverse Events (participants affected / at risk) | 30/65
Other Adverse Events (participants affected / at risk) | 62/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nab-paclitaxel and Ramucirumab (N=65)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3)
Death (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (7)
Sepsis (Infections and infestations) | 5 (5)
Septic shock (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Influenza B virus test positive (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Intramedullary rod insertion (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nab-paclitaxel and Ramucirumab (N=65)
Anaemia (Blood and lymphatic system disorders) | 12 (33)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (4)
Leukopenia (Blood and lymphatic system disorders) | 8 (13)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 29 (94)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (10)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Deafness (Ear and labyrinth disorders) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1)
Eye discharge (Eye disorders) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1)
Periorbital oedema (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 13 (17)
Abdominal pain upper (Gastrointestinal disorders) | 8 (10)
Ascites (Gastrointestinal disorders) | 4 (4)
Cheilitis (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 11 (14)
Diarrhoea (Gastrointestinal disorders) | 13 (26)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Gingival ulceration (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (2)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Lip haemorrhage (Gastrointestinal disorders) | 1 (1)
Lip ulceration (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 17 (28)
Oesophageal pain (Gastrointestinal disorders) | 2 (2)
Oral dysaesthesia (Gastrointestinal disorders) | 2 (2)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 9 (11)
Toothache (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (18)
Asthenia (General disorders) | 6 (7)
Axillary pain (General disorders) | 1 (1)
Catheter site erythema (General disorders) | 2 (2)
Chest pain (General disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 29 (54)
Localised oedema (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 9 (16)
Non-cardiac chest pain (General disorders) | 1 (1)
Oedema (General disorders) | 2 (3)
Oedema peripheral (General disorders) | 14 (18)
Pain (General disorders) | 3 (3)
Performance status decreased (General disorders) | 1 (1)
Pyrexia (General disorders) | 7 (10)
Swelling face (General disorders) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Abscess oral (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Candida infection (Infections and infestations) | 3 (3)
Catheter site infection (Infections and infestations) | 4 (4)
Colonic abscess (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Fungal skin infection (Infections and infestations) | 2 (2)
Genital herpes (Infections and infestations) | 1 (1)
Genital herpes simplex (Infections and infestations) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1)
Herpes ophthalmic (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Nasal herpes (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 4 (4)
Oral herpes (Infections and infestations) | 1 (1)
Penile infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Septic shock (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Staphylococcal skin infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 5 (6)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (6)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Stoma site ulcer (Injury, poisoning and procedural complications) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 2 (5)
Blood alkaline phosphatase increased (Investigations) | 3 (7)
Blood bilirubin increased (Investigations) | 2 (2)
Blood folate decreased (Investigations) | 1 (1)
Blood iron decreased (Investigations) | 2 (2)
Blood magnesium decreased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Clostridium test positive (Investigations) | 1 (1)
Colonoscopy (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 8 (15)
Oesophagogastroduodenoscopy (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (3)
Quality of life decreased (Investigations) | 1 (1)
Weight decreased (Investigations) | 16 (20)
Weight increased (Investigations) | 2 (2)
White blood cell count decreased (Investigations) | 1 (2)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 24 (31)
Dehydration (Metabolism and nutrition disorders) | 13 (16)
Fluid retention (Metabolism and nutrition disorders) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (3)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (6)
Aphasia (Nervous system disorders) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)
Cluster headache (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 8 (8)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (6)
Neuropathy peripheral (Nervous system disorders) | 15 (30)
Paraesthesia (Nervous system disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 2 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (12)
Sensory loss (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Taste disorder (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Device malfunction (Product Issues) | 1 (1)
Device occlusion (Product Issues) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (5)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3)
Mental status changes (Psychiatric disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 9 (13)
Urinary retention (Renal and urinary disorders) | 2 (3)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 16 (17)
Blister (Skin and subcutaneous tissue disorders) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (1)
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 3 (3)
Nail disorder (Skin and subcutaneous tissue disorders) | 3 (3)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 4 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Abscess drainage (Surgical and medical procedures) | 1 (1)
Gastrostomy tube removal (Surgical and medical procedures) | 1 (1)
Incisional drainage (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 8 (16)
Hypotension (Vascular disorders) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT02317991/Prot_SAP_000.pdf